CLINICAL TRIAL: NCT02810496
Title: Prevalence of Mutations of Glucocorticoid Receptors in Bilateral Adrenal Hyperplasia
Brief Title: Mutations of Glucocorticoid Receptor in Bilateral Adrenal Hyperplasia
Acronym: MUTA-GR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PN11010
Record Dates: First submitted 2016-06-16; First posted 2016-06-23 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2024-08

CONDITIONS: General Glucocorticoid Resistance

ARMS (1):
- patient (Experimental)
  Interventions: Genetic: blood collection for mutation characterization

INTERVENTIONS:
Genetic: blood collection for mutation characterization

SUMMARY:
As the investigators observed a case of glucocorticoid mutation revealed by incidentally discovered bilateral adrenal nodular hyperplasia, it was postulated that this molecular anormality could be more frequent than previously described. To validate this hypothesis, it was decided to study 150 multicenter consecutive patients, presenting with incidentally discovered bilateral adrenal masses without clinical signs of Cushing's disease. In all these patients GR gene will be studied, mutations will be detected and described, functional disturbance will be tested. Usual polymorphisms will be described. Correlation between clinical signs, hormonal and morphological abnormalities and presence or absence of GR mutations will be searched.

ELIGIBILITY:
Inclusion Criteria:

* patients more than 18 years of age
* patients with bilateral adrenal masses

Exclusion Criteria:

* Refusing to participate in the study
* Protected by law
* Have obvious signs of Cushing's syndrome
* No progressive neoplastic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-04-02 (Actual); Primary Completion 2016-10-02 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
frequency of mutations | DAY 0

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

REFERENCES:
- [Background] Vitellius G, Delemer B, Caron P, Chabre O, Bouligand J, Pussard E, Trabado S, Lombes M. Impaired 11beta-Hydroxysteroid Dehydrogenase Type 2 in Glucocorticoid-Resistant Patients. J Clin Endocrinol Metab. 2019 Nov 1;104(11):5205-5216. doi: 10.1210/jc.2019-00800. PMID 31225872
- [Result] Vitellius G, Trabado S, Hoeffel C, Bouligand J, Bennet A, Castinetti F, Decoudier B, Guiochon-Mantel A, Lombes M, Delemer B; investigators of the MUTA-GR Study. Significant prevalence of NR3C1 mutations in incidentally discovered bilateral adrenal hyperplasia: results of the French MUTA-GR Study. Eur J Endocrinol. 2018 Apr;178(4):411-423. doi: 10.1530/EJE-17-1071. Epub 2018 Feb 14. PMID 29444898